CLINICAL TRIAL: NCT03801863
Title: The Use of Lumbar Erector Spinae Plane Block for Hip Arthroplasty at the L4 Interspace- a Randomized Controlled Study Comparing the 24-hour Opioid Requirements.
Brief Title: The Use of Lumbar Erector Spinae Plane Block for Hip Arthroplasty at the L4 Interspace
Status: Terminated | Type: Observational
Why Stopped: Study "Administratively closed" by Albert Einstein College of Medicine IRB as approval expired. PI no longer with institution. IRB approval expiry date used as Primary Completion date and Study Completion Date. Enrollment total derived from CTMS
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-9687
Record Dates: First submitted 2019-01-05; First posted 2019-01-14 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Hip Arthropathy; Regional Anesthesia
Keywords: Erector Spinae Plane Block; Ropivacaine; Ultrasound guided nerve block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ultrasound-guided Erector Spinae Block: Patients will then be randomized into one of the two groups above. One group will receive a lumbar erector spinae block at L4 with 30ml of 0.375% ropivacaine with 50 mcg of dexmedetomidine before the procedure using ultrasound guidance. The second group will receive no peripheral nerve block to serve as the control. All patients receiving nerve blocks will have a printed image of the block thus to confirm proper spread of local anesthetic both cranially and caudally.
  Interventions: Procedure: Ultrasound-guided Erector Spinae Plane Block with Ropivacaine 0.375%; Drug: Ropivacaine
- No Ultrasound-guided Erector Spinae Block: Patients with no peripheral nerve block to serve as the control.

INTERVENTIONS:
Procedure: Ultrasound-guided Erector Spinae Plane Block with Ropivacaine 0.375% — Ultrasound-guided Erector Spinae Plane Block will be done at L4 interspace. Ropivacaine 0.375% will be used.
  Groups: Ultrasound-guided Erector Spinae Block
Drug: Ropivacaine — Using 0.375% Ropivacaine in the nerve block
  Groups: Ultrasound-guided Erector Spinae Block

SUMMARY:
Over 300,000 hip arthroplasties are performed each year in the United States.1 This number has been steadily increasing over the last two decades, likely due to increased life expectancy and, more significantly, the obesity epidemic. Traditionally, this procedure has been performed under general anesthesia. However, neuraxial and regional anesthesia have become more commonly utilized to aid in postoperative analgesia. Postoperative pain control has a significant impact on earlier ambulation, initiation of physical therapy, better functional recovery, and overall patient satisfaction.2 Moreover; optimal pain management can reduce the duration of hospitalization and the risk of adverse events, such as deep vein thrombus. The use of regional anesthesia reduces the postoperative opioid requirement, thereby decreasing the degree to which patients suffer the side effects of opioids, namely sedation and constipation, and less frequently nausea, vomiting, respiratory depression, pruritus, and retention. In the past, femoral nerve block, fascia iliaca compartment block, lumbar plexus block and the quadratus lumborum block have been shown efficacious for pain relief for hip arthroplasty. However there are several risk factors such as quadricep weakness and difficulty of the block that causes a limitation in the used of this blocks. Recently, the erector spinae plane block has been introduced as an alternative to the blocks above. This block was first described in the literature in 2016 when it was used to treat chronic neuropathic thoracic pain. Since then, there have been studies demonstrating its efficacy with a thoracic approach for analgesia in breast surgery and rib fractures.9 Only two case reports to date have demonstrated a lumbar approach to achieve analgesia for hip arthroplasty.10,11 The purpose of the study is to determine whether or not a lumbar erector spinae plane block is effective at improving postoperative pain in patients receiving hip arthroplasty.

DETAILED DESCRIPTION:
Hypothesis:

The erector spinae plane block will decrease opioid requirements in patients undergoing hip arthroplasty as compared to patients that do not receive the block.

Primary Objective:

To compare the opioid consumption in the post-anesthesia care unit (PACU) and at 24 hours postoperative (in morphine equivalents) in patients receiving regional anesthesia with spinal vs. spinal alone.

Secondary Endpoints:

To evaluate the pain scores at discharge from PACU, at 2 hours post PACU discharge, at 24 hours and at 48 hours postoperative; to evaluate the sensory distribution of the block (T10-L5); to evaluate whether or not patients that receive the block have evidence of quadricep muscle weakness

Design and methods This is a randomized, prospective study in patients receiving hip arthroplasty. Patients will be assigned to receive a lumbar erector spinae block versus no block. There will be no change in the primary anesthetic technique (spinal anesthesia with sedation) since these patients routinely get spinal anesthesia for hip arthroplasty. Consent for the study will be obtained in the preoperative area upon arrival for surgery. Patients will then be randomized into one of the two groups above. One group will receive a lumbar erector spinae block at L4 with 30ml of 0.375% ropivacaine with 50 mcg of dexmedetomidine before the procedure using ultrasound guidance. The second group will receive no peripheral nerve block to serve as the control. Patients to receive a nerve block will receive mild sedation (1-2mg midazolam ± ≤100mcg fentanyl). All patients receiving nerve blocks will have a printed image of the block thus to confirm proper spread of local anesthetic both cranially and caudally.

Postoperatively, the PACU nurse will be asked to document pain scores according to the Visual Analog Scale (VAS) and total dose of opioids given. The distribution of the sensory block and motor weakness will be documented in the anesthesiologist's PACU discharge note. For patients that receive the block, the Physical therapist note will be assessed for any report of quadriceps muscle weakness (i.e., evidence of buckling while walking).

For postoperative data collection, opioid consumption totals and the pain scores at 2 hours post admission, at 24 hours and 48 hours post-procedure will be collected from the electronic medical record (EMR) as documented by nurses on the admitting floor. Additionally, the Acute Pain service, who rounds on all patients that receive nerve blocks, will make a note of the pain scores of the patient and any residual muscle weakness or decreased sensation at 24- and 48-hours post-procedure. All data will then be extracted from the EMR by the research assistant.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary hip arthroplasty
* American Society of Anesthesiologists (ASA) Category 1, 2, and 3
* Patients age ≥18 years

Exclusion Criteria:

* Patient refusal
* Inability to understand and sign consent
* Infection at the injection site
* Known allergy or hypersensitivity to ropivacaine or other amide local anesthetics
* Contraindication or patient refusal to get spinal anesthesia
* Thrombocytopenia (platelets < 100,000)
* Coagulopathy (INR > 1.4)
* Use of anticoagulant drugs that have not been discontinued in an appropriate amount of time before the surgery
* ASA Category 4 and 5

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary total hip replacement under neuraxial anesthesia
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption in PACU and 24 hours post surgery | 24 hours
  To compare the opioid consumption in the post-anesthesia care unit (PACU) and at 24 hours postoperative (in morphine equivalents) in patients receiving regional anesthesia with spinal vs. spinal alone.

SECONDARY OUTCOMES:
Pain scores at 2 hours post PACU discharge | 2 hours. Pain scores from 1 to 10. 10 being the worse pain and 1 being the least pain
  To evaluate the pain scores at 2 hours post PACU discharge
To evaluate the sensory distribution of the block (T10-L5). | 2 hours post-surgery
  Will test for temperature difference using ice cube.
To evaluate whether or not patients that receive the block have evidence of quadricep muscle weakness | 30 hours post-surgery
  Will have patient walk and Physical Therapist will assess for buckling of knee or potential falls while ambulating.
Pain scores at 24 hours post PACU discharge | 24 hours. Pain scores from 1 to 10. 10 being the worse pain and 1 being the least pain
  To evaluate the pain scores at 24 hours post PACU discharge
Pain scores at 48 hours postoperative | 48 hours post-surgery. Pain scores from 1 to 10. 10 being the worse pain and 1 being the least pain
  To evaluate the pain scores at 48 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Iyabo Muse, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center- Wakefield Campus, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolford ML, Palso K, Bercovitz A. Hospitalization for total hip replacement among inpatients aged 45 and over: United States, 2000-2010. NCHS Data Brief. 2015 Feb;(186):1-8. PMID 25714040
- [Background] Bugada D, Bellini V, Lorini LF, Mariano ER. Update on Selective Regional Analgesia for Hip Surgery Patients. Anesthesiol Clin. 2018 Sep;36(3):403-415. doi: 10.1016/j.anclin.2018.04.001. Epub 2018 Jul 11. PMID 30092937
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005
- [Background] Tulgar S, Senturk O. Ultrasound guided Erector Spinae Plane block at L-4 transverse process level provides effective postoperative analgesia for total hip arthroplasty. J Clin Anesth. 2018 Feb;44:68. doi: 10.1016/j.jclinane.2017.11.006. Epub 2017 Nov 14. No abstract available. PMID 29149734
- [Background] Tulgar S, Selvi O, Senturk O, Ermis MN, Cubuk R, Ozer Z. Clinical experiences of ultrasound-guided lumbar erector spinae plane block for hip joint and proximal femur surgeries. J Clin Anesth. 2018 Jun;47:5-6. doi: 10.1016/j.jclinane.2018.02.014. Epub 2018 Mar 6. No abstract available. PMID 29522966
- [Background] Duellman TJ, Gaffigan C, Milbrandt JC, Allan DG. Multi-modal, pre-emptive analgesia decreases the length of hospital stay following total joint arthroplasty. Orthopedics. 2009 Mar;32(3):167. PMID 19309064